CLINICAL TRIAL: NCT04284722
Title: Perioperative Continuation of Metformin Therapy in Patients With Typ 2 Diabetes Mellitus Undergoing Non-cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Jens Meier, Prof. Jens Meier, MD, Kepler University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1126/2019
Record Dates: First submitted 2020-02-20; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Hyperglycemia; Metformin; Type 2 Diabetes; Hyperlactatemia
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus, Type 2; Hyperlactatemia | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin + (Active Comparator): The study intervention involves the self-administration of metformin in the same dosage as the patient's regular dosage according to regular dosing schedule and randomization.
  Interventions: Drug: Metformin Hydrochloride
- Metformin - (No Intervention): The control group involves no intervention, which means cessation of oral metformin therapy 24 hours prior to surgery according to the local guidelines of the anesthesia department and the national anesthesiology guidelines.

INTERVENTIONS:
Drug: Metformin Hydrochloride — Perioperative continuation of oral metformin therapy according to the patient's normal dosage and dosage intervals
  Other Names: Group A
  Arms: Metformin +

SUMMARY:
Evaluation of the effect of peri-operative continuation of oral metformin therapy on the incidence of perioperative hyperglycemia compared to standard preoperative cessation of oral metformin therapy 24h before surgery.

DETAILED DESCRIPTION:
Surgical procedures cause metabolic stress and can impair glucose control especially in patients with diabetes mellitus, which often results in peri-operative hyperglycemia. Peri-operative hyperglycemia is associated with impaired wound healing, secondary wound infections, endothelial dysfunction, sepsis, prolonged hospital stay and higher mortality.

Metformin is still the first line treatment in patients with type 2 diabetes mellitus.

Historically it has been stopped before surgery due to fear of hypoglycemia and metformin induced lactic acidosis. However recent studies have suggested that perioperative continuation of metformin might be safe and patients could benefit from more stable preoperative blood sugar levels.

Prospective studies evaluating the benefit of continuing oral metformin therapy in the perioperative period are rare.

The investigators plan to conduct a prospective, randomized-controlled, unblinded clinical trial where patients with type II diabetes mellitus and oral metformin therapy undergoing non-cardiac surgery will be randomized in either an interventional group or a control group. In the interventional group patients will be instructed to continue their regular metformin dose even on the day of surgery, in contrast to the control group, where the patients will be instructed to stop taking metformin 24h prior to surgery.

All other oral anti-diabetic drugs will be paused according to the local anesthesia guidelines.

The investigators plan to evaluate whether or not continuation of metformin can reduce the incidence of perioperative hyperglycemia and whether or not it is associated with elevation of blood lactate levels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99 years
* Diabetes Mellitus Typ 2
* Oral metformin therapy
* Non cardiac-surgery
* Informed consent

Exclusion Criteria:

* Insulin therapy
* Ambulatory surgery
* Preoperative therapy with glucocorticoids (prednisolon or equivalent ≥ 5mg/day for more than 7 days)
* Planned postoperative ICU-stay
* Advanced renal insufficiency (eGFR < 45ml/kg/min)
* Advanced liver cirrhosis or failure (Child-Pugh B or C)
* Alcohol abuse
* Pregnancy,
* Perioperative administration of contrast dye

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Perioperative Hyperglycemia | 24 hours pre-op until 24 hours post-op
  blood glucose >180mg/dl (10mmol/l) and/or necessity of additive administration of insulin s.c. during the time frame

SECONDARY OUTCOMES:
Perioperative blood glucose control | 24 hours pre-op until 24 hours post-op
  mean plasma glucose at 4 defined dates: 24h pre-op, intra-op, 2hours post-op and 24h post-op
Incidence hypoglycemia | 24 hours pre-op until 24 hours post-op
  blood sugar levels < 70mg/dl (3.9mmol/l)
Perioperative lactate levels | 24 hours pre-op until 24 hours post-op
  mediane lactate levels at 4 defined dates: 24h pre-op, intra-op, 2 hours post-op and 24h post-op
Incidence of hyperlactatemia | 24 hours pre-op until 24 hours post-op
  blood lactate values >4mmol/L at least at one of 4 measurement dates: 24h pre-op, intra-op, 2 hours post-op, 24 hours post-op
Perioperative renal function | 24 hours pre-op until 24 hours post-op
  median serum-creatinine value at 24h pre-op and 24h post-op
Hospitalization Duration | up to 4 weeks
  median time period from day of surgery until discharge from hospital
Mortality | up to 4 weeks
  In-Hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jens Meier, MD, Principal Investigator — Kepler University Hospital -Dpt. of Anesthesiology & Intensive Care Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hulst AH, Polderman JAW, Ouweneel E, Pijl AJ, Hollmann MW, DeVries JH, Preckel B, Hermanides J. Peri-operative continuation of metformin does not improve glycaemic control in patients with type 2 diabetes: A randomized controlled trial. Diabetes Obes Metab. 2018 Mar;20(3):749-752. doi: 10.1111/dom.13118. Epub 2017 Oct 13. PMID 28940961
- [Background] Gasanova I, Meng J, Minhajuddin A, Melikman E, Alexander JC, Joshi GP. Preoperative Continuation Versus Interruption of Oral Hypoglycemics in Type 2 Diabetic Patients Undergoing Ambulatory Surgery: A Randomized Controlled Trial. Anesth Analg. 2018 Oct;127(4):e54-e56. doi: 10.1213/ANE.0000000000003675. PMID 30044293
- [Background] Kuzulugil D, Papeix G, Luu J, Kerridge RK. Recent advances in diabetes treatments and their perioperative implications. Curr Opin Anaesthesiol. 2019 Jun;32(3):398-404. doi: 10.1097/ACO.0000000000000735. PMID 30958402
- [Background] Salpeter SR, Greyber E, Pasternak GA, Salpeter EE. Risk of fatal and nonfatal lactic acidosis with metformin use in type 2 diabetes mellitus. Cochrane Database Syst Rev. 2010 Apr 14;2010(4):CD002967. doi: 10.1002/14651858.CD002967.pub4. PMID 20393934